CLINICAL TRIAL: NCT07185932
Title: Efficacy and Safety of Rifaximin in Treating Metabolic Associated Fatty Liver Disease: A Pilot Trial
Brief Title: Efficacy and Safety of Rifaximin in Treating MAFLD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Department of Gastroenterology, Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZXH2021001.02
Record Dates: First submitted 2025-08-21; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Metabolic-associated Fatty Liver Disease
Keywords: metabolic-associated fatty liver disease; Rifaximin
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: Participants will receive oral rifaximin at a dosage of 1200 mg/day (400 mg, three times daily) for 24 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rifaximin treatment group (Experimental): Participants will receive oral rifaximin.
  Interventions: Drug: Rifaximin (Xifaxan)

INTERVENTIONS:
Drug: Rifaximin (Xifaxan) — Participants will receive oral rifaximin at a dosage of 1200 mg/day (400 mg, three times daily) for 24 weeks.

SUMMARY:
Study Objective: to evaluate the efficacy and safety of rifaximin in the treatment of metabolic-associated fatty liver disease (MAFLD), and investigate the underlying mechanisms by which rifaximin influence MAFLD progression.

Target Population: patients diagnosed with MAFLD. Intervention: this single-center, single-arm exploratory study will enroll up to 40 eligible MAFLD patients who meet the inclusion criteria, do not meet any exclusion criteria, and provide written informed consent. Participants will receive oral rifaximin at a dosage of 1200 mg/day (400 mg, three times daily) for 24 weeks. Patients will be advised to maintain their usual physical activity and adhere to a recommended dietary plan (e.g., Mediterranean diet). Concurrent therapies such as hepatoprotective agents, lipid-lowering medications, and antihypertensive treatments will remain unchanged, with close monitoring of relevant parameters. No additional prescription or over-the-counter drugs that may affect fatty liver progression or alter gut microbiota composition will be permitted during the study.

The primary endpoint will be assessed at 24 weeks. If liver proton density fat fraction (PDFF) remains ≥ 8% after 24 weeks of rifaximin therapy, treatment will be extended for an additional 12 weeks, followed by reevaluation of PDFF changes. The maximum total treatment duration will not exceed 48 weeks. All patients will undergo a 24-week post-treatment follow-up period after discontinuation of rifaximin.

Investigational Drug: Rifaximin (Alfa Wassermann S.p.A., Italy).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent;
2. Aged 18 to 75 years, regardless of gender;
3. Diagnosed with fatty liver disease within the past 6 months;
4. Presence of at least one of the following metabolic abnormalities:

(1) Overweight or obesity (BMI ≥23 kg/m²) (2) Type 2 diabetes (T2DM) (3) Clinical evidence of metabolic dysfunction (defined as meeting at least two of the following criteria): A. Waist circumference ≥90 cm for males or ≥80 cm for females B. Blood pressure ≥130/85 mmHg and/or diagnosed hypertension under treatment C. Fasting plasma triglycerides ≥1.7 mmol/L (150 mg/dL) or diagnosed hypertriglyceridemia under treatment D. Fasting HDL-C <1.0 mmol/L (40 mg/dL) for males or <1.3 mmol/L (50 mg/dL) for females, or diagnosed dyslipidemia under treatment E. Prediabetes: fasting glucose 5.6-6.9 mmol/L (100-125 mg/dL) or 2-hour postprandial glucose 7.8-11.0 mmol/L (140-199 mg/dL) or HbA1c 5.7%-6.4% (39-47 mmol/mol) F. Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) score ≥2.5 G. Plasma high-sensitivity C-reactive protein (hs-CRP) >2 mg/L 5. Liver fat content ≥8% as measured by MRI proton density fat fraction (MRI-PDFF).

Exclusion Criteria

1. Cirrhosis - Confirmed by clinical, laboratory, imaging, and/or liver biopsy.
2. Chronic liver disease of other etiologies (e.g., viral/autoimmune hepatitis, alcoholic liver disease, drug-induced liver injury)
3. Secondary hepatic steatosis (e.g., drug-induced, total parenteral nutrition-related, or hypothyroidism-associated);
4. Recent use of intestinal flora-modifying agents, or unstable regimens of medications (including hepatoprotectants, metformin, thiazolidinediones, fibrates, statins, et al) within 4 weeks prior to enrollment;
5. Agents with potential effects on MAFLD progression administered within 12 weeks prior to enrollment, excluding those maintained at stable doses for ≥24 weeks (e.g., Glucagon-like peptide-1 receptor agonists, Dipeptidyl peptidase IV inhibitors, Obeticholic acid, Sodium-glucose cotransporter 2 inhibitors, Resmetirom or anti-obesity medications)
6. Poorly controlled diabetes (HbA1c >9%)
7. Jaundice (total bilirubin ≥85 μmol/L), or Renal dysfunction (serum creatinine ≥1.2 × ULN)
8. History of bariatric surgery
9. Active or suspected malignancy
10. Severe systemic conditions - Including: Inflammatory diseases (e.g., connective tissue disorders), Biliary/pancreatic disorders, Chronic/acute infections, Severe cardiovascular, pulmonary, or hematologic diseases, Myocardial infarction or stroke within 6 months, Psychiatric disorders
11. HIV infection
12. Known hypersensitivity to rifaximin
13. MRI contraindications - Including: Metal implants, Claustrophobia, Body size exceeding scanner capacity
14. Pregnancy, lactation, or planned pregnancy
15. Participation in another drug trial within 3 months
16. Other conditions deemed unsuitable by investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in liver fat content measured by MRI at 24 weeks of treatment. | From enrollment to the end of treatment at 24 weeks
  Absolute and relative changes in MRI-measured liver proton density fat fraction (PDFF) at 24 weeks compared to baseline.

SECONDARY OUTCOMES:
Proportion of patients achieving ≥30% reduction in liver fat content measured by MRI-PDFF at 24 weeks of treatment compared to baseline | From enrollment to the end of treatment at 24 weeks
  Proportion of patients achieving ≥30% reduction in liver fat content measured by MRI-PDFF at 24 weeks of treatment compared to baseline
The change in liver fat content measured by MRI-PDFF at 12 weeks of treatment. | From enrollment to the end of treatment at 24 weeks
  Absolute and relative changes in MRI-measured liver PDFF at 12 weeks compared to baseline.
Proportion of patients achieving ≥30% reduction in liver fat content (PDFF) measured by MRI at 12 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 24 weeks
  The proportion of patients whose liver fat content (PDFF), assessed via MRI, decreased by ≥30% from baseline after 12 weeks of treatment.
Changes in liver function indicators after 12 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 weeks
  Changes in liver function parameters from baseline after 12 weeks of treatment.
Changes in liver function indicators after 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 24 weeks
  Changes in liver function indicators after 24 weeks of treatment compared to baseline.
Change in liver fat content assessed via FibroScan after 12 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 weeks
  Change in controlled attenuation parameter (CAP) values, measured by FibroScan, from baseline after 12 weeks of therapy
Change in liver fat content assessed via FibroScan after 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 24 weeks
  Change in controlled attenuation parameter (CAP) values, measured by FibroScan, from baseline after 24 weeks of therapy
Changes in fatty liver index (FLI) after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  FLI is utilized to assess the severity of hepatic steatosis. Its calculation formula is based on laboratory and anthropometric measurements, including triglyceride (TG) and gamma-glutamyl transferase (GGT) levels, body mass index (BMI), and waist circumference (WC).
  FLI = (e^(0.953 * ln(triglycerides) + 0.139 * BMI + 0.718 * ln(ggt) + 0.053 * waist circumference - 15.745)) / (1 + e^(0.953 * ln(triglycerides) + 0.139 * BMI + 0.718 * ln(ggt) + 0.053 * waist circumference - 15.745)) * 100
  A FLI value below 30 can be used to rule out steatosis (sensitivity = 87%; negative likelihood ratio [LR-] = 0.2), while a FLI value equal to or above 60 can be used to rule in hepatic steatosis.
Changes in NAFLD-liver fatty score（NAFLD-LFS）after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  NAFLD-LFS Calculation Formula: NAFLD-LFS = -2.89 + 0.45 × Type 2 Diabetes (yes=2, no=0) + 1.18 × Metabolic Syndrome (yes=1, no=0) + 0.15 × Insulin (mU/L) + 0.04 × AST (U/L) - 0.94 × (AST/ALT Ratio).
  Interpretation of Scores:
  NAFLD-LFS < -1.0: Suggests low liver fat content and a low likelihood of significant steatosis. -1.0 ≤ NAFLD-LFS ≤ 0.5: Intermediate range; further evaluation with additional tests (e.g., imaging or biopsy) is recommended. NAFLD-LFS > 0.5: Indicates high liver fat content and the presence of significant steatosis, requiring clinical intervention.
Changes in AST-to-Platelet Ratio Index (APRI) after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  APRI is calculated using the following formula:
  APRI = [ (AST Level (U/L) / AST ULN (Upper Limit of Normal)) / Platelet Count (10⁹/L) ] × 100
  Interpretation:
  APRI < 0.5: Suggests the absence of significant fibrosis (high negative predictive value).
  APRI > 2.0: Highly indicative of cirrhosis (high positive predictive value). Intermediate values (0.5 ≤ APRI ≤ 2.0): Further evaluation with additional tests-such as liver elastography, FIB-4 index, or liver biopsy-is recommended for accurate assessment.
Changes in Fibrosis 4 (FIB-4) Score after 12 and 24 weeks of treatment | From enrollment to the end of treatment at 12 and 24 weeks
  The FIB-4 index is primarily used to stratify the risk of liver fibrosis and is calculated using the following formula: FIB-4= Age (years) × AST (U/L)/ [Platelet Count (10⁹/L)×√ALT(U/L)]. The criteria are categorized as follows: Low Risk (FIB-4 < 1.3) suggests minimal or no fibrosis (F0-F1). Liver biopsy or elastography may be deferred in such cases. Intermediate Risk (1.3 ≤ FIB-4 ≤ 2.67): Further evaluation with additional tests-such as liver elastography, APRI, or liver biopsy-is recommended. Significant fibrosis (F2-F3) may be present, warranting closer monitoring. High Risk (FIB-4 > 2.67): Highly suggestive of advanced fibrosis or cirrhosis (F3-F4). Confirmatory tests like elastography or liver biopsy should be prioritized. This range has a high positive predictive value.
Changes in NAFLD fibrosis score (NFS) after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  NFS calculation formula: NFS= [-1.675+0.037×Age (years)+0.094×BMI（kg/m2+1.13×IFG/Diabetes (yes = 1, no = 0) +0.99）× (AST/ALT Ratio) +0.013×PLT(×109/L)-0.66×ALB（g/dl）]
  Interpretation Guidelines:
  NFS < -1.455: Low probability of significant fibrosis (F2-F4). NFS > 0.676: High probability of advanced fibrosis (F3-F4). NFS between -1.455 and 0.676: Indeterminate range; further evaluation with additional tests (e.g., elastography or liver biopsy) is recommended.
Changes in FibroScan-AST (FAST) Score after 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  The FAST Score is a non-invasive composite index used to assess the likelihood of both significant fibrosis (≥F2) and active steatohepatitis (NASH) in patients withMASLD. It integrates Liver Stiffness Measurement (LSM) obtained via FibroScan® and the serum biomarker AST.
  FAST Score Calculation Formula: FAST = e^(-1.65 + 1.07 × ln(LSM) + 2.66 × 10^(-8) × AST^3 - 63.3 × AST^(-1) - 0.009 × PLT) / (1 + e^(-1.65 + 1.07 × ln(LSM) + 2.66 × 10^(-8) × AST^3 - 63.3 × AST^(-1) - 0.009 × PLT)).
  Interpretation Guidelines:
  FAST < 0.35: Low probability of significant fibrosis (≥F2) with active inflammation (NASH). Negative predictive value >90%. Liver biopsy may be avoided.
  FAST > 0.67: High probability of both significant fibrosis (≥F2) and active inflammation (NASH). Positive predictive value >70%. Further evaluation or intervention is recommended.
  FAST between 0.35-0.67: Gray zone; comprehensive assessment with additional methods.
Changes in Body Mass Index (BMI) at 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  BMI calculation Formula:
  BMI = Weight (kilograms) ÷ [Height (meters)]²
Changes in Waist circumference (WC) at 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  Waist circumference (WC) is measured 3 cm above the navel.
Changes in visceral adipose tissue (VAT) at 12 and 24 weeks of treatment compared to baseline. | From enrollment to the end of treatment at 12 and 24 weeks
  VAT was quantified using 3D Slicer software by manually segmenting regions of interest (ROIs) within the intra-abdominal cavity on MRI images at the level of the third lumbar vertebra (L3).
Changes in abdominal subcutaneous adipose tissue (ASAT) from baseline after 12 and 24 weeks of therapy. | From enrollment to the end of treatment at 12 and 24 weeks
  ASAT volume was quantified using 3D Slicer software by manually segmenting regions of interest (ROIs) within the subcutaneous fat compartment on MRI images at the level of the third lumbar vertebra (L3).
Changes in Cholesterol from baseline after 12 and 24 weeks of therapy. | From enrollment to the end of treatment at 12 and 24 weeks
  Cholesterol testing should be performed in the morning after an overnight fast.
Changes in triglyceride from baseline after 12 and 24 weeks of therapy. | From enrollment to the end of treatment at 12 and 24 weeks
  Triglyceride testing should be performed in the morning after an overnight fast.
Changes in Hemoglobin A1c (HbA1c) from baseline after 12 and 24 weeks of therapy. | From enrollment to the end of treatment at 12 and 24 weeks
  Change from baseline in HbA1c absolute concentration (mmol/mol) and percentage of total hemoglobin (%) after 12 and 24 weeks of therapy.
Changes in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) from baseline after 12 and 24 weeks of therapy. | From enrollment to the end of treatment at 12 and 24 weeks
  HOMA-IR Calculation Formula: HOMA-IR = [Fasting Insulin (μIU/mL) × Fasting Glucose (mmol/L)] / 22.5. Increase in HOMA-IR suggests worsening insulin resistance. Decrease in HOMA-IR indicates improved insulin sensitivity.
The frequency and severity of treatment-related adverse events (AEs) as assessed by CTCAE 5.0. | From enrollment to the end of treatment at 24 weeks
  The safety assessment involved monitoring changes in symptoms, vital signs, and laboratory parameters during treatment.

OTHER OUTCOMES:
Changes in liver fat content assessed via MRI-PDFF during extended treatment (36 or 48 weeks) and at 12/24 weeks post-treatment. | Through study completion, an average of 3 years
  Longitudinal changes in liver PDFF measured by MRI during extended therapy (36 or 48 weeks) and after treatment discontinuation (12 and 24 weeks post-treatment), compared to baseline values

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng Hospital, Naval Medical University, shanghai, China, Shanghai, Shanghai Municipality, China